CLINICAL TRIAL: NCT03253159
Title: Added Conversational Hypnosis Reduced General Anesthesia Side Effects for Day Case Breast Surgery: A Prospective Randomized Phase III Clinical Trial (HYPNOSEIN)
Brief Title: Added Conversational Hypnosis Reduced General Anesthesia Side Effects for Day Case Breast Surgery
Acronym: HYPNOSEIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ICM-URC-2014/30
Record Dates: First submitted 2016-08-29; First posted 2017-08-17 (Actual); Last update posted 2020-08-10 (Actual); Status verified 2020-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Hypnosis

STUDY DESIGN:
Intervention Model Description: Hypnosis before intravenous anesthesia versus no preparation before intravenous anesthesia
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hypnosis group (Experimental): The conversational hypnosis (10-15 min) is standardized and performed just before intravenous general anesthesia induction in the operative room
  Interventions: Behavioral: Hypnosis
- Control group (No Intervention): No special preparation before intravenous general anesthesia induction in the operative room

INTERVENTIONS:
Behavioral: Hypnosis — The conversational hypnosis (10-15 min) is standardized and performed just before intravenous general anesthesia induction in the operative room.
  Arms: Hypnosis group

SUMMARY:
Evaluate the impact of the support in reducing postoperative adverse events in particular on the pain but also on anxiety, comfort, nausea, vomiting, and fatigue.

DETAILED DESCRIPTION:
Drug premedication with anxiolytics (benzodiazepine or equivalent) are usually prescribed to alleviate patient anxiety. However, alternative techniques, additional non-pharmacological, have proven effective in alleviating pain and anxiety perioperative. These techniques are retained relaxation therapy, reinsurance, breathing techniques and medical hypnosis as a technique of choice. Regarding medical hypnosis techniques, many studies have shown that performing a hypnotic technique performed perioperative could reduce the doses of anesthetics, postoperative pain, length of stay in the post room Interventional (SSPI) and a number of postoperative adverse effects.

Among the various techniques of hypnosis that can be offered to patients in the perioperative, conversational hypnosis is to accompany the patient on admission to the block to realization of general anesthesia. This technique aims to suggest a pleasant environment and not anxiety.

This study evaluate the impact of this support in reducing postoperative major adverse effects in particular on the pain but also on anxiety, comfort, nausea, vomiting, and fatigue.

ELIGIBILITY:
Inclusion Criteria:

* Female > 18 years
* Patient with ASA* score 1, 2, 3
* Minor Unilateral breast surgery indication (tumorectomy, lumpectomy, limited axillary node dissection, minor breast reconstruction…)
* Day case surgery (ambulatory surgery - living Day0-Day1)
* General anesthesia required
* Written informed consent
* French medical benefit

Exclusion Criteria:

* Age < 18 years
* Patient with ASA score > 4;
* Body mass index < 15 or 45kg/T;
* Major Surgery indication : mastectomy, bilateral surgery, full axillary dissection, major breast reconstruction
* Patient refusing hypnosis
* Psychic or mental Disorders
* Chronic pain
* Opiate therapeutic > 3 months
* Not ability to speak and read French language
* Deaf and dumb patient
* Under guardianship patient or guardianship

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2017-02-22 (Actual)

PRIMARY OUTCOMES:
Assessment of pain scale | through study completion, an average of 5 year
  Pain intensity assessment

SECONDARY OUTCOMES:
Reduction of the pain using Visual Analogic Scale | through study completion, an average of 5 year
  Reduction of the pain adverse postoperative outcome:
  Using Visual Analogic Scale (VAS > 3/10)

CONTACTS AND LOCATIONS:
Overall Officials: jibba AMRAOUI, Study Chair — Institut régional du Cancer de Montpellier
Locations (1):
- Institut réginal du Cancer de Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Amraoui J, Pouliquen C, Fraisse J, Dubourdieu J, Rey Dit Guzer S, Leclerc G, de Forges H, Jarlier M, Gutowski M, Bleuse JP, Janiszewski C, Diaz J, Cuvillon P. Effects of a Hypnosis Session Before General Anesthesia on Postoperative Outcomes in Patients Who Underwent Minor Breast Cancer Surgery: The HYPNOSEIN Randomized Clinical Trial. JAMA Netw Open. 2018 Aug 3;1(4):e181164. doi: 10.1001/jamanetworkopen.2018.1164. PMID 30646110